CLINICAL TRIAL: NCT03220763
Title: Eating Away from Home and Subsequent Risk of All-cause Mortality in the US Population
Brief Title: Eating Away from Home and Risk of All-cause Mortality
Status: Completed | Type: Observational
Sponsor: Queens College, The City University of New York (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ashima Kant, Professor, Queens College, The City University of New York
Other Study IDs: 69741-00 47; 69741-00 47 (Other Grant/Funding Number: PSC-CUNY)
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2019-03

CONDITIONS: Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thirds of number of restaurant meals: Respondent self-reports of # of times/week restaurant prepared meals were consumed. The respondents will be categorized into approximate thirds.
  Interventions: Other: This is an observational study--there is no intervention.

INTERVENTIONS:
Other: This is an observational study--there is no intervention. — This is an observational study, there is no intervention.

SUMMARY:
The proposed study will test the hypothesis that frequency of eating away from home meals is independently related to the prospective risk of mortality in the US population. The study will use public-domain mortality linked data from US national Surveys to address this question.

DETAILED DESCRIPTION:
This study uses public domain data collected in the National Health and Nutrition Examination Surveys (NHANES) conducted in 1999-2000, 2001-2002, and 2003-2004 by the National Center for Health Statistics. Data on frequency of eating restaurant meals were collected at that time. The surveys have been linked to the National Death Index and mortality status information is available in public-release files. The investigators aim to examine if exposure to restaurant meals at baseline is prospectively linked to the risk of mortality. All data are anonymized and available in the public domain.

ELIGIBILITY:
Inclusion Criteria:

* National Health and Nutrition Examination Surveys, 1999-2004, respondent
* Aged 40 or older at baseline

Exclusion Criteria:

* Pregnant or lactating
* No mobile examination center exam
* No exposure information
* No National Death Index linkage
* No followup time

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are the original respondents of the National Health and Nutrition Examination Surveys conducted in 1999-2004. The surveys include a nationally representative sample of the US, non-institutionalized population.
Sampling Method: Probability Sample
Enrollment: 9107 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Through end date of National Death Index followup, 12/31/2011
  Mortality from all causes

SECONDARY OUTCOMES:
Cause-specific mortality | Through end date of National Death Index followup, 12/31/2011
  mortality from specific causes

CONTACTS AND LOCATIONS:
Overall Officials: Ashima Kant, PhD, Principal Investigator — Faculty at Queens College of CUNY

IPD SHARING:
Plan to Share IPD: No